CLINICAL TRIAL: NCT02731937
Title: Clinical Evaluation of a Dual Energy CT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 106-2015-GES-0005
Record Dates: First submitted 2016-03-24; First posted 2016-04-08 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: General CT Imaging
MeSH Terms: interventions — Tomography Scanners, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- GE Healthcare CT Revolution (CT scanner) (Other): Each subject will be scanned twice: the first time will be the subjects' clinically indicated CT exam and the second scan will be performed on the GE Healthcare CT Revolution (CT scanner) both scans will will be obtained.
  Interventions: Device: GE Healthcare Revolution CT Scanner (CT Scanner)

INTERVENTIONS:
Device: GE Healthcare Revolution CT Scanner (CT Scanner) — Raw CT Scan Data
  Other Names: CT scanner

SUMMARY:
The main purpose of this study is to collect clinical raw scan data and Scanner user feedback using dual energy CT (computed tomography) scan modes on the investigational CT scanner. Additionally, image quality using prototype reconstruction algorithms that are in development will be evaluated and compared to standard-of-care images acquired with regulatory cleared diagnostic CT scanners for feasibility assessment and engineering development. Compared to standard clinical single energy (kilovolt,kV) scanning, dual energy (kV) scanning s provides more information about the material composition of the scanned patient and may allow for improved tissue, tumor characterization, and improved image quality.

ELIGIBILITY:
Inclusion Criteria:

1. Who are 18 year of age or older;
2. Able to sign and date the informed consent form; AND
3. Who have in the past year undergone a clinically-indicated CT exam of the head, neck, chest, abdomen, pelvis, or extremities

Exclusion Criteria:

1. Who are pregnant or lactating;
2. Who were previously enrolled in this study;
3. For contrast-enhanced CT exams, anyone with known or suspected allergy to iodinated contrast agents;
4. For contrast-enhanced CT exams, anyone with known or suspected renal insufficiency as determined by site medical personnel;
5. Who are in need of urgent or emergent care;
6. Diabetic patients on metformin (Glucophage)
7. Who have any conditions that, in the opinion of the PI or designee, would interfere with the evaluation of the results or constitute a health hazard for the subject; AND
8. Who are unwilling to have GEHC personnel present for the CT exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Raw CT Scan Data | 3 months
  No outcome assessment is currently planned. Up to 60 subjects will be scanned using GE Healthcare's Revolution CT scanner for future engineering and regulatory purposes.

SECONDARY OUTCOMES:
Image Quality assessment | 3 months
  Likert Scale to assess image quality

CONTACTS AND LOCATIONS:
Overall Officials: Ali Islam, MD, Principal Investigator — St. Joseph's Helathcare

IPD SHARING:
Plan to Share IPD: No